CLINICAL TRIAL: NCT06785649
Title: The Effect of Lavender Herbal Tea on the Mental Health of Individuals With Misophonia: A Randomized Clinical Trial
Brief Title: The Efficacy of Lavender Herbal Tea in Misophonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-1-2024-SK
Record Dates: First submitted 2025-01-04; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Misophonia; Misophonia Treatment; Anxiety; Depression; Anger; Complementary Medicine
Keywords: misophonia; anxiety; depression; anger; lavender
MeSH Terms: conditions — misophonia; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The waiting list group, which is the control group, will not undergo any intervention. The experimental group will use lavender herbal tea in the morning and evening for 14 days.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (lavender herbal tea) (Experimental): Each participant will be allocated 14 pieces of lavender tea bags of 2 grams, originating from Turkey. The intervention group will be advised to use 2 g of lavender herb infused in 300 mL hot water for 10-15 minutes in the morning and evening for 14 days. Participants will be advised to take some time and inhale the scent before drinking the herbal tea.
  Interventions: Other: Lavender herbal tea
- Control group (wait-list) (No Intervention): No intervention will be applied to the control group for 14 days.

INTERVENTIONS:
Other: Lavender herbal tea — The participant will be allocated 14 pieces of lavender tea bags consisting of 2 grams and originating from Turkey. During 14 days, the participant will be advised to use 2 g of lavender herb brewed in 300 mL hot water for 10-15 minutes in the morning and evening. Participants will be able to use 1 lavender tea bag twice a day.
  Arms: Experimental group (lavender herbal tea)

SUMMARY:
Misophonia is a disorder characterized by a high level of annoyance with certain sounds. Exposure to these sounds causes physical symptoms characterized by anger, aggression, helplessness, overwhelm, and stimulation of the sympathetic nervous system. These emotional and physical reactions can lead to a decline in family relationships, work and school productivity, withdrawal from social relationships, and even suicide. There is limited empirical evidence evaluating the efficacy of therapeutic approaches to misophonia. This limited empirical evidence consists of pharmacological agents such as selective serotonin reuptake inhibitors, stimulants, antipsychotics, and β-Blockers, as well as cognitive behavioral therapy, acceptance and commitment therapy, and dialectical behavior therapy. Complementary therapies are important because of their potential efficacy, tolerability, possible non-interference, and low cost. The fact that lavender has anxiolytic, antidepressant, neuroprotective, and anti-inflammatory properties may affect the emotional and physical responses elicited by misophonia. Therefore, within the scope of the study, misophonia individuals will be divided into two groups; one group will use lavender tea for 14 days and the other group will form a waiting list. The study data will be collected by 'Information Collection Form', 'Misophonia Scale', 'Beck Depression Inventory-II', 'Anxiety Rating Scale', and 'Trait Anger Scale'. SPSS 25.0 software will be used to analyze the data obtained from the research. Considering the limitations of therapeutic approaches for misophonia, testing the effectiveness of lavender in reducing misophonia symptoms will make an important contribution to the literature.

DETAILED DESCRIPTION:
Misophonia is a disorder of vocal sensitivity characterized by unusual discomfort with certain sounds. Typical triggers are sounds produced by humans, particularly oral and nasal sounds. These sounds include chewing, slurping, breathing, keyboard sounds, or pen clicks. When individuals with misophonia are exposed to triggers, stimulation of the sympathetic nervous system and emotional distress are observed. Exposure to triggers creates irritation, desire to avoid stimuli, anger, aggression, helplessness, and overwhelm. Stimulation of the sympathetic nervous system leads to physical symptoms such as hypertonia, sweating, and tachycardia. The discomfort and stress caused by misophonia can lead to increased anxiety levels in individuals. At the same time, the emotional distress and discomfort associated with misophonia can trigger depressive symptoms and increase the risk of depression. Concomitant anxiety and depression can worsen the existing symptoms of misophonia and lead to a reduced quality of life.

There is limited empirical evidence evaluating the efficacy of therapeutic approaches to misophonia. Current treatment approaches include cognitive behavioral therapy, acceptance and commitment therapy, and psychotherapies derived from dialectical behavior therapy. Due to the small number of randomized controlled trials, the efficacy of the protocols used in the treatment of misophonia remains unclear. Due to limited resources, problems such as limited access to psychotherapies and early withdrawal from treatment are also observed. Other treatment approaches include pharmacological agents such as selective serotonin reuptake inhibitors (SSRIs), stimulants, antipsychotics, and β-Blockers. Complementary therapies are used due to their potential efficacy, tolerability, possible non-interference, and low cost. Lavender, a complementary treatment intervention, is considered to have anxiolytic, antidepressant, neuroprotective, and anti-inflammatory properties. Lavender is known to positively affect memory, provide alertness, and improve feelings of well-being. Thus, it is seen as an effective herbal medicine intervention in reducing anxiety and depression. Reducing concomitant anxiety and depression may contribute to the improvement of the symptoms of misophonia.

ELIGIBILITY:
Inclusion Criteria:

* Reporting at least three trigger sounds
* Assessed by a specialist psychiatric nurse and a psychiatrist as humophonia based on the diagnostic criteria for humophonia established by Schröder et al. (2013)
* Individuals aged 18 and over

Exclusion Criteria:

* Allergy to any herbal tea, food or medicine
* Psychiatric illness or chronic illness
* Taking psychiatric medication (such as anxiolytics, and antidepressants)
* Regular use of medication (such as antihypertensive, antidiabetic)
* Regular use of herbal teas or complementary medicines
* Tinnitus and/or hyperacusis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Misophonia Scale | Within the first 24 hours after 14 days of lavender tea
  It is a 30-item self-report scale aiming to assess the severity of misophonia. The scale is a 5-point Likert-type scale and is graded between 1: Strongly agree and 5: Strongly disagree to 5: Strongly disagree. The total score range is 30 - 150. As the score obtained from the scale decreases, the level of misophonia severity decreases.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Within the first 24 hours after 14 days of lavender tea
  It is a 21-item self-report inventory aimed at assessing the severity of depression. The items are rated from 0 to 3 depending on the severity of symptoms. The total score range is 0 to 63 and is divided into four grades in terms of severity: minimal depression (total score 0-13), mild depression (14-19), moderate depression (20-28) and severe depression (≥ 29).
Anxiety Assessment Scale | Within the first 24 hours after 14 days of lavender tea
  This scale, which evaluates anxiety, consists of 10 items. The scale is in 5-point Likert type and is expressed as 1: Never, 2: Very Rarely, 3: Sometimes, 4: Often, 5: Almost Always. There are no reverse scored items in the scale, the total scale score of anxiety is obtained by summing all items. The lowest score that can be obtained from the scale is 10 and the highest score is 50. The higher the total score, the higher the level of anxiety.
Trait Anger Scale (SL-Anger) | Within the first 24 hours after 14 days of lavender tea
  This scale is an assessment tool that measures how often and at what level individuals feel anger in their lives. Consisting of 10 items, this test is graded with a four-point Likert type (1=Never, 2=Sometimes, 3=Most of the time, 4=Always). The increase in the total score obtained from the scale indicates that the individual tends to feel anger more frequently and more intensely in his/her life.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kianpour M, Moshirenia F, Kheirabadi G, Asghari G, Dehghani A, Dehghani-Tafti A. The Effects of Inhalation Aromatherapy with Rose and Lavender at Week 38 and Postpartum Period on Postpartum Depression in High-risk Women Referred to Selected Health Centers of Yazd, Iran in 2015. Iran J Nurs Midwifery Res. 2018 Sep-Oct;23(5):395-401. doi: 10.4103/ijnmr.IJNMR_116_16. PMID 30186346
- [Background] Firoozeei TS, Feizi A, Rezaeizadeh H, Zargaran A, Roohafza HR, Karimi M. The antidepressant effects of lavender (Lavandula angustifolia Mill.): A systematic review and meta-analysis of randomized controlled clinical trials. Complement Ther Med. 2021 Jun;59:102679. doi: 10.1016/j.ctim.2021.102679. Epub 2021 Feb 4. PMID 33549687
- [Background] Su S, Wang Y, Jiang W, Zhao W, Gao R, Wu Y, Tao J, Su Y, Zhang J, Li K, Zhang Z, Zhao M, Wang Z, Luo Y, Huang X, Wang L, Wang X, Li Y, Jia Q, Wang L, Li H, Huang J, Qiu J, Xu Y. Efficacy of Artificial Intelligence-Assisted Psychotherapy in Patients With Anxiety Disorders: A Prospective, National Multicenter Randomized Controlled Trial Protocol. Front Psychiatry. 2022 Jan 20;12:799917. doi: 10.3389/fpsyt.2021.799917. eCollection 2021. PMID 35126211
- [Background] Rappoldt LR, van der Pol MM, de Wit C, Slaghekke S, Houben C, Sondaar T, Kan KJ, van Steensel FJAB, Denys D, Vulink NCC, Utens EMWJ. Effectiveness of an innovative treatment protocol for misophonia in children and adolescents: Design of a randomized controlled trial. Contemp Clin Trials Commun. 2023 Mar 11;33:101105. doi: 10.1016/j.conctc.2023.101105. eCollection 2023 Jun. PMID 36950304
- [Background] Jager IJ, Vulink NCC, Bergfeld IO, van Loon AJJM, Denys DAJP. Cognitive behavioral therapy for misophonia: A randomized clinical trial. Depress Anxiety. 2020 Dec 18;38(7):708-18. doi: 10.1002/da.23127. Online ahead of print. PMID 33336858
- [Background] Cowan, E. N., Marks, D. R., & Pinto, A. Misophonia: A psychological model and proposed treatment. Journal of Obsessive-Compulsive and Related Disorders, 32, 100691. https://doi.org/10.1016/j.jocrd.2021.100691
- [Background] Jager I, de Koning P, Bost T, Denys D, Vulink N. Misophonia: Phenomenology, comorbidity and demographics in a large sample. PLoS One. 2020 Apr 15;15(4):e0231390. doi: 10.1371/journal.pone.0231390. eCollection 2020. PMID 32294104
- [Background] Cassiello-Robbins C, Anand D, McMahon K, Brout J, Kelley L, Rosenthal MZ. A Preliminary Investigation of the Association Between Misophonia and Symptoms of Psychopathology and Personality Disorders. Front Psychol. 2021 Jan 14;11:519681. doi: 10.3389/fpsyg.2020.519681. eCollection 2020. PMID 33519567
- [Background] Erfanian M, Kartsonaki C, Keshavarz A. Misophonia and comorbid psychiatric symptoms: a preliminary study of clinical findings. Nord J Psychiatry. 2019 May-Jul;73(4-5):219-228. doi: 10.1080/08039488.2019.1609086. Epub 2019 May 8. PMID 31066600
- [Background] Brout JJ, Edelstein M, Erfanian M, Mannino M, Miller LJ, Rouw R, Kumar S, Rosenthal MZ. Investigating Misophonia: A Review of the Empirical Literature, Clinical Implications, and a Research Agenda. Front Neurosci. 2018 Feb 7;12:36. doi: 10.3389/fnins.2018.00036. eCollection 2018. PMID 29467604
- [Background] Swedo SE, Baguley DM, Denys D, Dixon LJ, Erfanian M, Fioretti A, Jastreboff PJ, Kumar S, Rosenthal MZ, Rouw R, Schiller D, Simner J, Storch EA, Taylor S, Werff KRV, Altimus CM, Raver SM. Consensus Definition of Misophonia: A Delphi Study. Front Neurosci. 2022 Mar 17;16:841816. doi: 10.3389/fnins.2022.841816. eCollection 2022. PMID 35368272
- [Derived] Koroglu Gokbel S, Durat G. The effect of lavender herbal tea on the mental health of individuals with misophonia: A randomized controlled trial. J Psychiatr Res. 2026 Jan 21;195:39-46. doi: 10.1016/j.jpsychires.2026.01.028. Online ahead of print. PMID 41579454